CLINICAL TRIAL: NCT03436147
Title: Vaginally Assisted Laparoscopic Hysteropexy Versus Vaginal Hysterectomy for the Treatment of Uterovaginal Prolapse: a Prospective Randomized Study
Brief Title: Vaginally Assisted Laparoscopic Hysteropexy Versus Vaginal Hysterectomy
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ismail Alay, principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: VALHvsVAH
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: vaginal hysterectomy; laparoscopic hysteropexy; pelvic organ prolapse quantification
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaginal Assisted Laparoscopic Sacrohysteropexy(VALH): Patients who were performed vaginal assisted laparoscopic sacrohysteropexy (VALH)
  Interventions: Other: POP-Q
- Vaginal Hysterectomy and Vaginal vault suspension (VAH+VVS): Patients who were performed vaginal hysterectomy and vaginal vault suspension(VAH+VVS)
  Interventions: Other: POP-Q

INTERVENTIONS:
Other: POP-Q — Pelvic Organ Prolapse Quantification

SUMMARY:
Utero-vaginal prolapse is a common, often disabling, condition experienced by women of varying ages. The traditional surgical treatment for utero-vaginal prolapse often includes vaginal hysterectomy and anterior or posterior colporrhaphy. Growing emphasis on patient-centered medicine and patient-generated definitions of surgical success has resulted in reassessment of uterine preservation versus hysterectomy at the time of apical POP repair. Various techniques have been described for uterine preserving prolapse surgery, which may include vaginal sacrospinous hysteropexy, transvaginal mesh kits, abdominal sacrohysteropexy using mesh and laparoscopic uterine suspension using sling or mesh. A modified form of uterine-preserving prolapse surgery using a combined vaginal and laparoscopic approach was introduced and a series of 70 women was reported. To date, there have been no randomized studies comparing the outcomes of vaginal assisted laparoscopic uterine suspension (hysteropexy) with conventional vaginal hysterectomy. Women attending the gynecology clinic at a tertiary referral urogynecology unit in tertiary referral training and research hospital requesting surgical treatment for STAGE 2-4 symptomatic uterine prolapse will be offered participation in a randomized trial, over a 2-year period. Subjects participating in the study were randomly assigned to either of two groups: Group A, Vaginally Assisted Laparoscopic Hysteropexy (VALH), or Group B, Vaginal Hysterectomy and Mc Call Culdoplasty (VH + Mc Call).1 year following surgery, vaginal prolapse will be assessed again using the International Consultation on Incontinence Questionnaire for Vaginal Symptoms (ICIQ-VS) questionnaire and the Pelvic Organ Prolapse -Quantification (POP-Q) examination by another researcher then the operator.

DETAILED DESCRIPTION:
Utero-vaginal prolapse is a common, often disabling, condition experienced by women of varying ages. The traditional surgical treatment for utero-vaginal prolapse often includes vaginal hysterectomy and anterior or posterior colporrhaphy. Growing emphasis on patient-centered medicine and patient-generated definitions of surgical success has resulted in reassessment of uterine preservation versus hysterectomy at the time of apical pelvic organ prolapse (POP) repair. Comparison of study outcomes between hysteropexy and hysterectomy are confounded by anatomic variables (isolated apical prolapse or multiple compartment prolapse), hormonal status (premenopausal, postmenopausal on hormone therapy, and postmenopausal without hormone therapy), and surgical approach (vaginal, open abdominal, laparoscopic, and robotic). In addition, the number of women who subsequently undergo hysterectomy after a uterus-sparing prolapse surgery is not known. With the caveat of these limitations, new short-term data are available to inform consideration of uterine-sparing POP repair. Various techniques have been described for uterine preserving prolapse surgery, which may include vaginal sacrospinous hysteropexy, transvaginal mesh kits, abdominal sacrohysteropexy using mesh and laparoscopic uterine suspension using sling or mesh. A modified form of uterine-preserving prolapse surgery using a combined vaginal and laparoscopic approach was introduced and a series of 70 women was reported.To date, there have been no randomized studies comparing the outcomes of vaginal assisted laparoscopic uterine suspension (hysteropexy) with conventional vaginal hysterectomy.

This is a single-center, randomized controlled study of two parallel groups. Women attending the gynecology clinic at a tertiary referral urogynecology unit requesting surgical treatment for STAGE 2-4 symptomatic uterine prolapse will be offered participation in a randomized trial, over a 2-year period between February 2018 and February 2020.

Requirements for women recruited are that

* patients who are over 35 years of age with no desire to preserve fertility. (Subjects had completed childbearing or were practicing reliable contraception)
* have a normal size uterus (<10 cm) on examination or ultrasound
* who agree to participate in principle will be given further information about the trial and consent will be obtained either in an outpatient clinic or at the next visit for preoperative assessment.

Investigators will exclude women with

* cervical elongation (surgeon discretion),
* prior mesh prolapse repair,
* current foreign-body complications,
* increased risk or recent history of cervical dysplasia, chronic pelvic pain, significant uterine abnormalities, and abnormal menstruation.
* Postmenopausal bleeding in the past 12 months
* Women with a significantly enlarged fibroid uterus or concomitant medical problems precluding general anesthesia or the use of a steep Trendelenburg position Subjects participating in the study will be randomly assigned to either of two groups: Group A, Vaginally Assisted Laparoscopic Hysteropexy (VALH), or Group B, Vaginal Hysterectomy and Vaginal Vault Suspension (VAH + VVS). Those recruited who subsequently have a strong preference or either operation and consequently decline to continue in the study will be excluded and will not randomized.

VALH surgical procedure described below:

The procedure was performed under general anesthesia with the patient initially in the lithotomy position. After insertion of a urinary catheter, a 2 cm transverse vaginal incision was performed to the posterior cervix. The vaginal mucosa on the posterior cervix was dissected and type 1 polypropylene mesh secured to the posterior cervix with six 2/0 polydioxanone sutures. After skin preparation, and draping, a pneumoperitoneum was created and three laparoscopic ports were placed; 11 mm umbilical, 5 mm left and right lateral ports, and 5 mm suprapubic port. The sacral promontory was subsequently visualized and the presacral peritoneum was opened with monopolar diathermy and laparoscopic scissors.The tail end of the mesh was then push forward to the promontorium in the retroperitoneal region under laparoscopic visualisation. The end of the mesh grasped and pulled up laparoscopically. The uterus pushed up to the using the uterine manipulator. The mesh was then tacked to the sacral promontory with 5 mm helical fasteners. Finally, the mesh was completely covered with peritoneum, gas was expelled and ports were withdrawn under vision. Skin incisions were closed with absorbable fine sutures.

On the day of the operation allocation will be confirmed and appropriate consent will be obtained for the specific surgical procedure. Vaginal hysterectomy + Mc Call Culdoplasty and vaginal assisted laparoscopic hysteropexy will combined with anterior and/or posterior repair depending on the judgment of the surgeon at the time of the operation. Each woman will be followed up initially in the clinic 3 months post-surgery as part of the departmental routine. Participants will then invite for review, as part of the trial, at a dedicated clinic, 1 year following surgery. Vaginal prolapse will be assessed again using the International Consultation on Incontinence Questionnaire for Vaginal Symptoms (ICIQ-VS) questionnaire and the Pelvic Organ Prolapse Quantification (POP-Q) examination by another researcher then the operator. During the interview, further questions will be asked regarding post-operative recovery, current urinary symptoms, Urogenital Distress Inventory Short Form (UDI-6) and the Incontinence Impact Questionnaire Short Form (IIQ-7) and their satisfaction with the operation. Subjective surgical outcome will be measured using the Patient Global Impression of Improvement (PGI-I), which is a validated tool as a global index of response to prolapse surgery.

The women's prolapse symptoms and their impact will be evaluated before surgical treatment.

1. A subjective assessment of the prolapse will be made using the ICIQ-VS
2. Objective assessment of pelvic organ prolapse will be performed during a Valsalva maneuver, in the left lateral position, using a Sims' speculum. Investigators use the pelvic organ prolapse quantification (POP-Q) system.
3. Patients will be also asked to complete the Urogenital Distress Inventory Short Form (UDI-6) and the Incontinence Impact Questionnaire Short Form (IIQ-7). UDI-6 and IIQ-7 are accepted as validated questionnaires that are useful in the assessment of urogenital symptoms and disease-specific QoL.

The measure for primary outcome is treatment failure defined as recurrent apical prolapse surgery required within the first year post-operatively.

The secondary outcome measures are change in anatomy quantified by POP-Q and symptoms quantified using the ICIQ-VS questionnaire scores for prolapse, sexual wellbeing, quality of life, and PGI-I score, UDI-6 and IIQ-7 scores. Other secondary outcome measures are operation time, blood loss, hospital stay, and time before return to normal activity.

ELIGIBILITY:
Inclusion Criteria:

* patients who are over 35 years of age with no desire to preserve fertility. (Subjects had completed childbearing or were practicing reliable contraception)
* have a normal size uterus (<10 cm) on examination or ultrasound
* who agree to participate in principle will be given further information about the trial and consent will be obtained either in an outpatient clinic or at the next visit for preoperative assessment.

Exclusion Criteria:

* cervical elongation (surgeon discretion),
* prior mesh prolapse repair,
* current foreign-body complications,
* increased risk or recent history of cervical dysplasia, chronic pelvic pain, significant uterine abnormalities, and abnormal menstruation.
* postmenopausal bleeding in the past 12 months
* women with a significantly enlarged fibroid uterus
* concomitant medical problems precluding general anesthesia or the use of a steep trendelenberg position

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women attending the gynecology clinic at a tertiary referral urogynecology unit in our hospital requesting surgical treatment for STAGE 2-4 symptomatic uterine prolapse.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Kaya, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaginal Hysterectomy and Vaginal Vault Suspension(VAH+VVS): Patients who were performed a vaginal hysterectomy and Vaginal vault suspension
Period: Overall Study
Arm/Group | Vaginal Assisted Laparoscopic Sacrohysteropexy(VALH) | Vaginal Hysterectomy and Vaginal Vault Suspension(VAH+VVS)
Started | 19 | 30
Completed | 15 | 19
Not Completed | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Vaginal Hysterectomy and Vaginal Vault Suspensio (VAH+VVS): Patients who were performed a vaginal hysterectomy and Vaginal Vault Suspension (VAH + VVS)
  POP-Q: Pelvic Organ Prolapse Quantification
- Total: Total of all reporting groups
Arm/Group | Vaginal Assisted Laparoscopic Sacrohysteropexy(VALH) | Vaginal Hysterectomy and Vaginal Vault Suspensio (VAH+VVS) | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (9.1) | 64.0 (9.5) | 59.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 19 | 34
Region of Enrollment [Number; unit: participants]
  Turkey | 15 | 19 | 34
International Consultation on Incontinence Questionnaire Vaginal Symptoms (ICIQ-VS) [Mean (Standard Deviation); unit: units on a scale] — International Consultation on Incontinence Questionnaire-Vaginal Symptoms (ıcıq-vs ) score of the patient after postoperative one year. This score includes 14 questions as Dragging abdominal pain, Vaginal soreness, Reduced sensation around vagina, Vagina too loose/lax, Lump coming down in vagina, Lump coming out of vagina, Dry vagina, Digitation for bowel opening, Tight vagina, Current sex life, Worries about vagina affect sex life, Relationship Sex life spoilt, Overall impact on everyday life. ICIQ-VS score ranges between 0 and 53. Higher ICIQ-VS scores represent worse outcome.
  units on a scale | 20.9 (7.6) | 22.6 (6.2) | 21.8 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Pelvic Organ Prolapse
Description: Number of Participants with Recurrence of Pelvic Organ Prolapse
Time Frame: Postoperative first year
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Assisted Laparoscopic Sacrohysteropexy(VALH) | Vaginal Hysterectomy and Vaginal Vault Suspension (VAH+VVS)
Number analyzed (Participants) | 15 | 19
Participants | 0 | 0

2. Secondary Outcome: POP-Q SYSTEM Point C MEASUREMENT
Description: The POP-Q system is an objective, site-specific system for describing and staging POP in women. The measurement is then taken of the distance from the point to the hymenal plane. Point C is defined as the most distal (ie, most dependent) edge of the cervix or the leading edge of the vaginal cuff (posthysterectomy). Preoperative and postoperative one year measurement of point C according to POP-Q system will be recorded and the change from preoperative measurement at postoperative first year is secondary outcome of this study.
Time Frame: change from preoperative measurement of pop-q point c at postoperative first year
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Vaginal Assisted Laparoscopic Sacrohysteropexy(VALS): Patients who were performed vaginal assisted laparoscopic sacrohysteropexy (VALH)
  POP-Q: Pelvic Organ Prolapse Quantification
- Vaginal Hysterectomy and Vaginal Vault Suspension(VAH+VVS): Patients who were performed vaginal hysterectomy and Vaginal vault suspension
  POP-Q: Pelvic Organ Prolapse Quantification
Arm/Group | Vaginal Assisted Laparoscopic Sacrohysteropexy(VALS) | Vaginal Hysterectomy and Vaginal Vault Suspension(VAH+VVS)
Number analyzed (Participants) | 15 | 19
centimeters | -8.5 (3.4) | -7 (3.2)

3. Secondary Outcome: ICIQ-VS Vaginal Symptom Subscale
Description: International Consultation on Incontinence Questionnaire-Vaginal Symptoms (ıcıq-vs ) score of the patient after postoperative one year. This score includes 14 questions as Dragging abdominal pain, Vaginal soreness, Reduced sensation around vagina, Vagina too loose/lax, Lump coming down in vagina, Lump coming out of vagina, Dry vagina, Digitation for bowel opening, Tight vagina, Current sex life, Worries about vagina affect sex life, Relationship Sex life spoilt, Overall impact on everyday life. ICIQ-VS score ranges between 0 and 53. Higher ICIQ-VS scores represent worse outcome.
Time Frame: change from preoperative ICIQ-VS vaginal symptom subscale score at postoperative first year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaginal Assisted Laparoscopic Sacrohysteropexy(VALS) | Vaginal Hysterectomy and Vaginal Vault Suspension(VAH+VVS)
Number analyzed (Participants) | 15 | 19
score on a scale | -13.8 (7.6) | 17.7 (5.4)

ADVERSE EVENTS:
Time Frame: 12 months
Description: there was no adverse event observed in both groups
Arm/Group | Vaginal Assisted Laparoscopic Sacrohysteropexy(VALS) | Vaginal Hysterectomy and Vaginal Vault Suspension(VAH+VVS)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 0/15 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT03436147/Prot_SAP_000.pdf